CLINICAL TRIAL: NCT00369187
Title: Study of a Large Protein Molecule Administered With Escalating Doses of Recombinant Human Hyaluronidase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HZ2-06-02
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2008-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: large protein molecule

SUMMARY:
This Phase IV, dose escalation, within-patient controlled study of pharmacokinetics (PK), safety and tolerability compares a single dose administration of a large protein molecule without recombinant human hyaluronidase (rHuPH20) to a single dose administration of the large molecule with escalating doses of rHuPH20. The study hypothesizes that an optimal dose of rHuPH20 will increase the bioavailability of large molecule drug administration.

DETAILED DESCRIPTION:
Sequential enrollment into four rHuPH20 dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age with RA treated with MTX who have been treated with:

   * co-injected large molecule protein for at least two cycles, and
   * have had stable disease with no symptom flares in the previous 30 days.
2. AST (SGOT) and ALT (SGPT) within normal range within 7 days prior to entry in the study.
3. Adequate venous access in at least one extremity.
4. A negative pregnancy test (if female of child-bearing potential) within 7 days prior to entry in the study.
5. Decision-making capacity.
6. Signed, written IRB-approved informed consent.

Exclusion Criteria:

1. Unacceptable toxicity to the large molecule protein, or contraindication to or other reason to not continue the large molecule protein per the package insert (e.g., active or latent tuberculosis, chronic or localized infections, or concurrent treatment with anakinra).
2. History of active tuberculosis, or known positive tuberculin skin test unless the patient has successfully completed a nine-month course of isoniazid therapy.
3. Concurrent use of any disease-modifying anti-rheumatic drug except the large molecule protein and MTX.
4. Any anticipation that the dose of the large molecule protein or MTX would be changed within 4 weeks following entry in the study.
5. Known allergy to hyaluronidase or any hyaluronidase product.
6. Known allergy to bee or vespid venom.
7. Contraindication to IV heparin lock or known hypersensitivity to heparin.
8. Edema, infection, or any other lower extremity or pelvic disorder that might affect subcutaneous absorption from the thigh.
9. Presence of any other medical condition that would present an unacceptable safety risk to the patient.
10. Participation in a study of any investigational drug or device within 30 days of enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
AUC

SECONDARY OUTCOMES:
Tmax, Cmax, half-lives, injection site reactions, safety and tolerability, NAbs

CONTACTS AND LOCATIONS:
Overall Officials: Malin Prupas, M.D., Principal Investigator — Arthritic Center of Reno